CLINICAL TRIAL: NCT00325013
Title: Evaluation of Docosahexaenoic Acid (DHA) for the Treatment of Primary Sclerosing Cholangitis (PSC)
Brief Title: Evaluation of DHA for the Treatment of PSC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Steven Freedman, MD PhD Professor of Medicine at Harvard School of Medicine, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005P-000259 (DK71851); R03DK071851 (NIH)
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Primary Sclerosing Cholangitis; Colitis
Keywords: Primary Sclerosing Cholangitis; PSC; DHA; Docosahexaenoic Acid
MeSH Terms: conditions — Cholangitis, Sclerosing; Colitis | interventions — Docosahexaenoic Acids; Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- II (Experimental)
  Interventions: Drug: Docosahexaenoic Acid (DHA)

INTERVENTIONS:
Drug: Docosahexaenoic Acid (DHA) — 800mg twice a day for 1 year
  Other Names: fish oil

SUMMARY:
The researches aim to study the effects of DHA (component of fish oil) on patients with Primary Sclerosing Cholangitis (PSC). Our hypothesis is that DHA might reverse the problems associated with PSC.

DETAILED DESCRIPTION:
The etiology of Primary Sclerosing Cholangitis (PSC) is unknown. There are no proven effective therapies and no early markers of the disease to predict which patients with colitis may be at risk to develop PSC.

Our group has demonstrated an increased prevalence of CFTR alleles (the gene responsible for Cystic Fibrosis (CF)) in patients with PSC which was correlated with decreased CFTR function as measured by Nasal Potential Difference Testing. These data suggested that colitis in the setting of CFTR dysfunction may lead to bile duct inflammation and fibrosis. As proof of concept, we subsequently demonstrated in cftr-/- mice that (1) colitis leads to the development of bile duct injury and (2) this is prevented by correction of the CFTR related fatty acid defect with oral Docosahexaenoic Acid (DHA). Preliminary data in these mice indicates that low PPAR expression in the liver may predispose to inflammation. One mechanism by which DHA ameliorates the innate inflammatory response linked to CFTR dysfunction may be through an increase in PPAR expression.

Based on these data, we hypothesize that CFTR dysfunction may contribute to the pathogenesis of primary sclerosing cholangitis (PSC). Furthermore, correction of the fatty acid abnormality and changes in the innate immune response associated with CFTR dysfunction by oral administration of docosahexaenoic acid (DHA), an n-3 polyunsaturated fatty acid, might be an effective therapy for patients with PSC.

Immediate Objectives:

To evaluate the effect of DHA therapy on patients with PSC, examining:

Primary Outcome:

• serum alkaline phosphatase

Secondary Outcomes:

* cholangiography
* liver biochemistry (ALT, AST, gamma-glutamyl transferase, bilirubin, albumin, prothrombin time,)
* fatty acid profile (docosahexaenoic acid, arachidonic acid)
* serum/plasma liver fibrosis markers (hyaluronic acid, tumor necrosis factor-α, transforming growth factor-ß, type III procollagen peptide)
* innate immune response (peripheral blood monocytes for assessment of cytokine secretion, lipoxins, and PPAR)
* clinical data on signs and symptoms

ELIGIBILITY:
Inclusion Criteria:

Patients must have a diagnosis of primary sclerosing cholangitis. The diagnosis will require a chronic cholestatic liver disease of at least 6 months' duration; a serum alkaline phosphatase level at least 1.5 times the upper limit of normal; cholangiographic findings of intrahepatic or extrahepatic biliary-duct obstruction, beading, or narrowing consistent with PSC; and a liver biopsy in the previous 12 months with compatible findings.

Exclusion Criteria:

Age less than18 years or more than 80 years. Subjects must have no evidence of secondary cholangitis or other liver disease (primary biliary cirrhosis, alcoholic liver disease, autoimmune hepatitis, and chronic viral hepatitis). Subjects will be excluded if there is a history of previous bile duct surgery, previous choledocholithiasis, recurrent ascending cholangitis, previous history of variceal hemorrhage, or cholangiocarcinoma. Subjects with PSC stage III (fibrosis) or IV (cirrhosis) based on the criteria of Ludwig et al. will be excluded.

Participants will be excluded if there are pregnant.

Subjects will also be excluded if treatment with corticosteroids, cyclosporine or methotrexate has occurred within the preceding 3 months, or there is an anticipated need for liver transplantation within 1 year. No fish oil supplements will otherwise be allowed. Patients on 5-aminosalicylate preparations or azathioprine will remain on these preparations for the duration of the trial. Treatment with ursodeoxycholic acid will not be an exclusion criteria. Patients on this therapy will be advised to continue the drug throughout the trial. Those not on ursodeoxycholic acid will not be allowed to start this drug since it is could affect the alkaline phosphatase levels and is not an accepted efficacious therapy. Subjects will not be excluded for refusal of follow-up MRCP at study completion. There will be no exclusion based on sex, race, and ethnic background.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Primary outcome will be change in alkaline phosphatase. Outcome in alkaline phosphatase will be defined as:Highly positive: >50% reduction;Positive: >25% reduction; | 1 years
No Change: <25% reduction or <25% increase;Negative: >25% increase;Highly negative: >50% increase | 1 years

SECONDARY OUTCOMES:
Secondary outcomes will include changes in:cholangiography;liver biochemistry (ALT, AST, gamma-glutamyl transferase, bilirubin, albumin, prothrombin time);fatty acid profile (docosahexaenoic acid, arachidonic acid); | 1 years
serum/plasma liver fibrosis markers (hyaluronic acid, tumor necrosis factor-α, transforming growth factor-ß, type III procollagen peptide);peripheral blood monocyte PPAR (mRNA by RT-PCR, protein level by western blot, and activity by EMSA); | 1 year
peripheral blood monocyte cytokine secretion (IL-8) in response to Pseudomonas LPS, TNF, IL-10; lipoxin A4 secretion and lipoxygenase expression as well as docosatriene/resolvins;symptoms;safety measures of DHA (Adverse Event recordings) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Steve D Freedman, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota